CLINICAL TRIAL: NCT06742749
Title: Proximal Versus Distal Tenotomy of the Iliopsoas Tendon in the Surgical Treatment of Developmental Dysplasia of the Hip: a Randomized Clinical Trial
Brief Title: Level of Iliopsoas Tenotomy in DDH Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Duhok (Other)
Responsible Party: Principal Investigator, Jagar Omar Doski, Assistant Professor, University of Duhok
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Jagar Doski
Record Dates: First submitted 2024-12-14; First posted 2024-12-19 (Actual); Last update posted 2024-12-30 (Actual); Status verified 2024-12

CONDITIONS: Developmental Dysplasia of the Hip (DDH)
Keywords: Hip; Developmental Dysplasia of the hip; surgical treatment; Iliopsoas Tenotomy; Randomized Clinical Trial
MeSH Terms: conditions — Developmental Dysplasia of the Hip

STUDY DESIGN:
Intervention Model Description: The study was a randomized clinical trial. It was done to check the equivalence between two parallel groups of patients with DDH who underwent open reduction operation for their hips. In the first group, the psoas tendon was sectioned at the pelvic brim (proximal level), while in the second group, the section of the tendon was done just above the lesser trochanter (distal level). The allocation ratio was 1:1.
Who Masked: Participant, Outcomes Assessor
Masking Description: The patients, their parents/guardians, and the person who assessed the primary outcome were blinded to the type of intervention and the randomization sequence. The primary outcome assessor was a physiotherapist already trained in rehabilitating children with orthopedic disorders and the manual muscle strength testing scale. The assessment of the primary outcome was done in the physiotherapy department of the EDCD center.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group 1 (Experimental): For the proximal level of psoas tenotomy at the pelvic brim, the hip was slightly flexed to relax the iliopsoas muscle; the iliacus muscle fibers were retracted anteriorly until the deeply seated posteromedially psoas tendon was isolated and transected
  Interventions: Procedure: Proximal level
- Group 2 (Active Comparator): . For the distal level of iliopsoas tenotomy just above the lesser trochanter, the thigh was put in the position of FABER (flexion, abduction, and external rotation). A curved right-angle hemostatic clamp was used to retract and bring the iliopsoas tendon into the field. Then, the tendinous fibers were transected.
  Interventions: Procedure: Distal level

INTERVENTIONS:
Procedure: Proximal level — For the proximal level of psoas tenotomy at the pelvic brim, the hip was slightly flexed to relax the iliopsoas muscle; the iliacus muscle fibers were retracted anteriorly until the deeply seated posteromedially psoas tendon was isolated and transected
  Arms: Group 1
Procedure: Distal level — For the distal level of iliopsoas tenotomy just above the lesser trochanter, the thigh was put in the position of FABER (flexion, abduction, and external rotation). A curved right-angle hemostatic clamp was used to retract and bring the iliopsoas tendon into the field. Then, the tendinous fibers were transected.
  Arms: Group 2

SUMMARY:
The goal of this clinical trial is to compare the postoperative clinical outcome of iliopsoas tenotomy in open reduction operation for developmental dysplasia of the hip. The main aim is to compare the postoperative clinical outcome of division of iliopsoas tendon at two levels, proximally at the pelvic brim and distally just above the lesser trochanter.

DETAILED DESCRIPTION:
All the patients with DDH included in the current study underwent open reduction of their dislocated hip through the anterior approach. None of the included patients underwent hip surgery through the medial approach.

For the proximal level of psoas tenotomy at the pelvic brim, the hip was slightly flexed to relax the iliopsoas muscle; the iliacus muscle fibers were retracted anteriorly until the deeply seated posteromedially psoas tendon was isolated and transected. For the distal level of iliopsoas tenotomy just above the lesser trochanter, the thigh was put in the position of FABER (flexion, abduction, and external rotation). A curved right-angle hemostatic clamp was used to retract and bring the iliopsoas tendon into the field. Then, the tendinous fibers were transected.

ELIGIBILITY:
Inclusion Criteria:

* Children with DDH.
* Required open reduction of their hip problem.

Exclusion Criteria:

* Patients who underwent hip surgery without the need for sectioning the iliopsoas tendon.
* Children with mental retardation who were not cooperative in the assessment of the hip flexion strength.

Ages: 1 Year to 8 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 54 (Actual)
Dates: Start 2021-01-02 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2024-12-27 (Actual)

PRIMARY OUTCOMES:
hip flexion strength | at 6th, 12th, and 24th months post-operatively
  The strength was assessed clinically using the Medical Research Council Manual Muscle Testing scale. It evaluated muscle strength by testing the key muscle against gravity and the examiner's resistance. The scale graded muscle strength into six grades (from 0 to 5): Grade 0, no muscle activation and no movement; Grade 1, trace muscle activation, a flicker of movement, but without achieving full range of motion; Grade 2, muscle activation and achieving full range of motion with eliminated gravity; Grade 3, muscle activation and achieving full range of motion against gravity; Grade 4, muscle activation and achieving full range of motion against some resistance; Grade 5, muscle activation and achieving full range of motion against strong resistance.

SECONDARY OUTCOMES:
complications | 12 months
  : femoral nerve injury detected postoperatively by the inability to extend the knee actively from paralysis of the quadriceps muscle; medial circumflex femoral vessels injury detected intraoperatively by the active bleeding that may occur during iliopsoas tenotomy at the distal level (just above the lesser trochanter); avascular necrosis (AVN) of the femoral epiphysis detected postoperatively by the radiographic film when the femoral head failed to ossify or to grow within one year after being reduced, widening of the femoral neck within one year of reduction, changes in the bone density of the femoral head, and residual deformity that suggested growth disturbance

CONTACTS AND LOCATIONS:
Locations (1):
- College of Medicine/University of Duhok, Duhok, Iraq

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol
Time Frame: from 1 year till 5 years
Access Criteria: contact author